CLINICAL TRIAL: NCT00943202
Title: Effect of Administration of Licensed TIV Vaccine on the Safety and Immunogenicity of an Unadjuvanted Sanofi Pasteur H1N1 Influenza Vaccine in Previously Primed Infants and Toddlers (Greater Than or Equal to 6 - <36 Months), Children (Greater Than or Equal to 36 Months - 9 Years), and Adolescents (10 - 17 Years)
Brief Title: Sanofi Pasteur, TIV + H1N1, Pediatric Population
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 09-0047; N01AI80003C
Record Dates: First submitted 2009-07-21; First posted 2009-07-22 (Estimated); Results first posted 2011-05-26 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2010-12

CONDITIONS: Influenza
Keywords: H1N1, influenza A viruses, TIV, vaccine, infants, children
MeSH Terms: conditions — Influenza, Human

ARMS (4):
- Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV (Experimental): 150 subjects to receive-Day 0: 15 mcg H1N1 vaccine; Day 21: 15 mcg H1N1 vaccine; Day 42: TIV.
  Interventions: Biological: Inactivated H1N1 Vaccine; Biological: Trivalent Inactivated Influenza Vaccine
- Group 2: Day 0-H1N1+TIV; Day 21-H1N1 (Experimental): 150 subjects to receive-Day 0: 15 mcg H1N1 vaccine + TIV; Day 21: 15 mcg H1N1 vaccine.
  Interventions: Biological: Inactivated H1N1 Vaccine; Biological: Trivalent Inactivated Influenza Vaccine
- Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1 (Experimental): 150 subjects to receive-Day 0: TIV; Day 21: 15 mcg H1N1 vaccine; Day 42: 15 mcg H1N1 vaccine.
  Interventions: Biological: Inactivated H1N1 Vaccine; Biological: Trivalent Inactivated Influenza Vaccine
- Group 3: Day 0-H1N1; Day 21-H1N1+TIV (Experimental): 150 subjects to receive-Day 0: 15 mcg H1N1 vaccine; Day 21: 15 mcg H1N1 vaccine + TIV.
  Interventions: Biological: Inactivated H1N1 Vaccine; Biological: Trivalent Inactivated Influenza Vaccine

INTERVENTIONS:
Biological: Inactivated H1N1 Vaccine — Inactivated influenza H1N1 vaccine, 15 micrograms per dose. Vaccines will be administered as a single 0.5 mL intramuscular injection in the deltoid muscle of the arm or in the anterolateral thigh muscle (1 injection in each arm or each thigh if receiving 2 doses).
Biological: Trivalent Inactivated Influenza Vaccine — Licensed seasonal trivalent influenza vaccine (TIV) (2009-2010 season). For subjects greater than or equal to 6 - <36 months, licensed TIV will be administered as a single 0.25 mL intramuscular (IM) injection in the deltoid muscle of the arm or in the anterolateral thigh muscle. For subjects greater than or equal to 36 months - 17 years, licensed TIV will be administered as a single 0.5 mL IM injection in the deltoid muscle of the arm or in the anterolateral thigh muscle.

SUMMARY:
The purpose of this study is to assess the safety and immune response (body's defense against disease) to an experimental H1N1 influenza vaccine against the 2009 H1N1 virus. This study will help determine how and when the H1N1 flu shot should be given with the seasonal flu shot to make it most effective. The 650 participants will be divided into the following age groups: infants from 6 months-36 months old, children 36 months-9 years old, and adolescents 10-17 years old. Each age group will have 200 children. There are 4 treatment groups in each age level. Study procedures include: medical history, targeted physical exam based on history, maintaining a memory aid, and blood sample collection. Participants will be involved in the study for about 8 months.

DETAILED DESCRIPTION:
Recently, a novel swine-origin influenza A/H1N1 virus was identified as a significant cause of febrile respiratory illnesses in Mexico and the United States. It rapidly spread to many countries around the world, prompting the World Health Organization (WHO) to declare a pandemic on June 11, 2009. Data from several cohorts in different age groups that received licensed trivalent seasonal influenza vaccines suggest that these vaccines are unlikely to provide protection against the new virus. In addition, adults are more likely to have measurable levels of serum hemagglutination inhibition assay (HAI) or neutralizing antibody than are children. These data indicate the need to develop vaccines against the new H1N1 strain and suggest that different vaccine strategies (e.g., number of doses, need for adjuvant) may be appropriate for persons in different age groups. If the novel influenza H1N1 2009 virus continues to circulate, it is possible that it will co-circulate with the non-pandemic seasonal influenza strains. In this situation, it might be beneficial to co-administer an H1N1 vaccine concurrent with the seasonal inactivated influenza vaccine. This protocol will explore if vaccination with the 2009-2010 licensed seasonal trivalent influenza vaccine (TIV) has an effect on antibody response to the novel influenza H1N1 2009 virus. This protocol will also examine if receiving the H1N1 vaccine either concurrent with, prior to, or following the seasonal influenza vaccine affects the antibody response to the seasonal influenza vaccine. A randomized Phase II study in infants, toddlers, children and adolescents. This study is designed to investigate the safety, reactogenicity, and immunogenicity of an inactivated influenza H1N1 virus vaccine when given concurrent with seasonal TIV, or sequentially with (before or after) seasonal influenza vaccine. Primary objectives are: safety, to assess the safety of the unadjuvanted, inactivated H1N1 vaccine when administered either concurrent with, prior to, or following licensed seasonal influenza vaccination; and immunogenicity, to assess the effect of TIV administration on antibody response to unadjuvanted, inactivated H1N1 vaccine as assessed by HAI, stratified by age of recipient. The secondary objective is: immunogenicity, to assess the effect of H1N1 vaccine administration on antibody response to TIV as assessed by HAI, stratified by age of recipient. Subjects will be randomized into 4 groups, stratified by age (150 subjects per group with 50 subjects per age stratum: greater than or equal to 6-<36 months, greater than or equal to 36 months-9 years, and 10-17 years), to receive two 15 mcg doses of inactivated influenza H1N1 vaccine at Days 0 and 21 followed by TIV on Day 42 (Group 1), two 15 mcg doses of H1N1 vaccine of which the first dose is administered concurrently with TIV (Group 2), two 15 mcg doses of H1N1 vaccine of which the second dose is administered concurrently with TIV (Group 3), or TIV administered on Day 0 followed by two 15 mcg doses of H1N1 vaccine on Days 21 and 42 (Group 4). Following immunization, safety will be measured by assessment of adverse events for 21 days following the last vaccination (Day 42 for those who do not receive the second dose), serious adverse events and new-onset chronic medical conditions for 8 months post first vaccination (Day 201 for Groups 2 and 3 or Day 222 for Groups 1 and 4), and reactogenicity to the vaccines for 8 days following each vaccination (Day 0-7). Immunogenicity testing will include HAI and neutralizing antibody testing prior to vaccination, on the day of each vaccination (Days 0, 21 and 42) and 21 days following the third vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Are males or non-pregnant females aged 6 months to 17 years, inclusive.
* All subjects 6 months to 9 years must be "primed".
* Subjects of child-bearing potential must agree to practice adequate contraception that may include, but is not limited to, abstinence, barrier methods such as condoms, diaphragms, spermicides, intrauterine devices, and licensed hormonal methods during the study for at least 30 days following the last vaccination.
* The subject must be in good health, as determined by axillary (<10 years of age) or oral temperature (axillary temperature <100 degrees Fahrenheit or oral temperature <101 degrees Fahrenheit), medical history, and targeted physical examination based on medical history.
* Subject and/or parent(s)/legal guardian(s) must be willing and able to comply with planned study procedures and be available for all study visits.
* Subject and/or parent(s)/legal guardian(s) must provide written informed consent prior to initiation of any study procedures, and subject may provide written assent as appropriate.

Exclusion Criteria:

* Have a known allergy to eggs or other components of the vaccine (including gelatin, formaldehyde, octoxinol, thimerosal and chicken protein).
* Have a positive urine or serum pregnancy test within 24 hours prior to vaccination or are breastfeeding.
* Have immunosuppression as a result of an underlying illness or treatment, or use of anticancer chemotherapy or radiation therapy (cytotoxic) within the preceding 36 months.
* Have an active neoplastic disease or a history of any hematologic malignancy.
* Have long term use of glucocorticoids including oral, parenteral or high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) within the preceding 6 months. (Nasal and topical steroids are allowed.)
* Have a diagnosis of schizophrenia, bipolar disease, or other major psychiatric diagnosis or major depression.
* Have been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others.
* Are receiving any psychiatric drugs (aripiprazole, clozapine, ziprasidone, haloperidol, molindone, loxapine, thioridazine, thiothixene, pimozide, fluphenazine, risperidone, mesoridazine, quetiapine, trifluoperazine, chlorprothixene, chlorpromazine, perphenazine, trifluopromazine, olanzapine, carbamazepine, divalproex sodium, lithium carbonate or lithium citrate) or any drugs for treatment of depression.
* Have a history of receiving immunoglobulin or other blood product within the 3 months prior to vaccination in this study.
* Received an experimental agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month prior to vaccination in this study or expect to receive an experimental agent during the study period (prior to Day 180 after the last vaccination).
* Have received any live licensed vaccines within 4 weeks or inactivated licensed vaccines within 2 weeks prior to vaccination in this study or plan receipt of such vaccines within 21 days following the last vaccination. This is inclusive of routine childhood immunizations provided outside the scope of this study. The initiation of this protocol does not take precedence over routine immunizations.
* Has received a licensed 2009-2010 seasonal influenza vaccine.
* Have an acute or chronic medical condition that, in the opinion of the investigator, would render vaccination unsafe, or would interfere with the evaluation of responses.
* Have a history of severe reactions following previous immunization with influenza virus vaccines.
* Have an acute illness, including an axillary temperature greater than 100 degrees Fahrenheit or an oral temperature greater than or equal to 101 degrees Fahrenheit, within 3 days prior to vaccination.
* Have any condition that would, in the opinion of the site investigator, place them at an unacceptable risk of injury or render them unable to meet the requirements of the protocol.
* Participated in a novel influenza H1N1 2009 vaccine study in the past two years or have a history of novel influenza H1N1 2009 infection prior to enrollment.
* Have known active human immunodeficiency virus (HIV), Hepatitis B or Hepatitis C infection.
* Have a history of alcohol or drug abuse.
* Plan to travel outside of North America in the time between the first vaccination and 63 days following the first vaccination.
* Have a history of Guillain-Barré Syndrome.
* Have any condition that the investigator believes may interfere with successful completion of the study.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 531 (Actual)
Dates: Start 2009-08; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Emory Children's Center - Pediatric Infectious Diseases, Atlanta, Georgia
  - Emory University School of Medicine - Emory Children's Center - Pediatric Infectious Diseases, Atlanta, Georgia
  - University of Iowa, Iowa City, Iowa
  - Saint Louis University Hospital - Internal Medicine - Infectious Diseases, Allergy & Immunology, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Vanderbilt University - Pediatric - Vanderbilt Vaccine Research Center, Nashville, Tennessee
  - The University of Texas Medical Branch, Galveston, Texas
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Result] Frey SE, Bernstein DI, Gerber MA, Keyserling HL, Munoz FM, Winokur PL, Turley CB, Rupp RE, Hill H, Wolff M, Noah DL, Ross AC, Cress G, Belshe RB. Safety and immune responses in children after concurrent or sequential 2009 H1N1 and 2009-2010 seasonal trivalent influenza vaccinations. J Infect Dis. 2012 Sep 15;206(6):828-37. doi: 10.1093/infdis/jis445. Epub 2012 Jul 16. PMID 22802432
- [Derived] Kotloff KL, Halasa NB, Harrison CJ, Englund JA, Walter EB, King JC, Creech CB, Healy SA, Dolor RJ, Stephens I, Edwards KM, Noah DL, Hill H, Wolff M. Clinical and immune responses to inactivated influenza A(H1N1)pdm09 vaccine in children. Pediatr Infect Dis J. 2014 Aug;33(8):865-71. doi: 10.1097/INF.0000000000000329. PMID 25222307

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were healthy males and females, age 6 months to 17 years, recruited from existing volunteer populations and from the communities at large around the clinical sites. Participants were enrolled between 20AUG2009 and 21SEP2009.
Groups:
- Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV: Participants received 15 mcg H1N1 Vaccine on Day 0; 15 mcg H1N1 Vaccine on Day 21, and Trivalent Influenza Vaccine (TIV) on Day 42
- Group 2: Day 0-H1N1+TIV; Day 21-H1N1: Participants received 15 mcg H1N1 Vaccine + Trivalent Influenza Vaccine (TIV) on Day 0 and 15 mcg H1N1 Vaccine on Day 21
- Group 3: Day 0-H1N1; Day 21-H1N1+TIV: Participants received 15 mcg H1N1 Vaccine on Day 0 and 15 mcg H1N1 Vaccine + Trivalent Influenza Vaccine (TIV) on Day 21
- Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1: Participants received Trivalent Influenza Vaccine (TIV) on Day 0; 15 mcg H1N1 Vaccine on Day 21, and 15 mcg H1N1 Vaccine on Day 42.
Period: Overall Study
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Started | 133 | 133 | 133 | 132
Completed | 132 | 131 | 133 | 131
Not Completed | 1 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1 | Total
Number analyzed (Participants) | 133 | 133 | 133 | 132 | 531
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 133 | 133 | 133 | 132 | 531
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 8.0 (5.0) | 8.2 (5.3) | 7.9 (5.3) | 8.5 (5.0) | 8.1 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 71 | 57 | 57 | 253
  Male | 65 | 62 | 76 | 75 | 278
Region of Enrollment [Number; unit: participants]
  United States | 133 | 133 | 133 | 132 | 531

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Age 6 Months to Less Than 36 Months With 4-fold or Greater Hemagglutination Inhibition Assay (HAI) Antibody Titer Increases Against the Influenza H1N1 2009 Virus 21 Days Following the First Dose of H1N1 Vaccine
Description: Blood was collected from participants for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. A participant met the threshold of a 4-fold rise in titer if the Day 0 titer was less than 1:10 (the assay's lowest level of detection) and the Day 21 post first H1N1 vaccination titer was 1:40 or greater, or the Day 0 titer was greater than or equal to 1:10 and the Day 21 titer was an increase by 4-fold or more. Day 21 post first H1N1 vaccination is Study Day 42 for Group 4, and is Study Day 21 for all other groups.
Time Frame: Day 0 prior to vaccination and 21 days after the first H1N1 vaccination
Population: Participants who received the H1N1 vaccination and from whom blood was collected at the timepoint, both within 4 days of the window, are included. Analyses are as treated. This outcome restricts to age stratum.
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 35 | 30 | 33 | 26
Participants | 10 | 6 | 5 | 5

2. Primary Outcome: Number of Participants Age 36 Months to 9 Years With 4-fold or Greater Hemagglutination Inhibition Assay (HAI) Antibody Titer Increases Against the Influenza H1N1 2009 Virus 21 Days Following the First Dose of H1N1 Vaccine
Description: as for outcome 1
Time Frame: Day 0 prior to vaccination and 21 days after the first H1N1 vaccination
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 47 | 49 | 45 | 50
Participants | 20 | 21 | 19 | 20

3. Primary Outcome: Number of Participants Age 10 to 17 Years With 4-fold or Greater Hemagglutination Inhibition Assay (HAI) Antibody Titer Increases Against the Influenza H1N1 2009 Virus 21 Days Following the First Dose of H1N1 Vaccine
Description: as for outcome 1
Time Frame: Day 0 prior to vaccination and 21 days after the first H1N1 vaccination
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 49 | 48 | 46 | 51
Participants | 46 | 39 | 41 | 48

4. Primary Outcome: Number of Participants Age 6 to Less Than 36 Months Reporting Solicited Subjective Systemic Reactions After the First Vaccination
Description: Participants' parents/guardians maintained a memory aid to record daily the occurrence of systemic symptoms of irritability, decreased appetite and lethargy for 8 days after vaccination (Day 0-7) based on their interference with daily activities. Participants are counted if they were reported as experiencing the symptom at any severity on any of the 8 days.
Time Frame: Within 8 days (Day 0-7) post first vaccination
Population: All participants receiving the first vaccination are included in the safety cohort. Analyses are as treated. This outcome measure is restricted to protocol-defined age stratum.
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 35 | 33 | 35 | 28
Participants
  Irritability | 18 | 15 | 16 | 9
  Decreased appetite | 6 | 5 | 9 | 5
  Lethargy | 8 | 6 | 8 | 3

5. Secondary Outcome: Number of Participants Age 6 to Less Than 36 Months With 4-fold or Greater Hemagglutination Inhibition Assay (HAI) Antibody Titer Increases Against the Virus Strains in the 2009-2010 Trivalent Influenza Vaccine (TIV) 21 Days Following the Last Vaccination
Description: Blood was collected from participants for testing in the HAI assay against each strain in the 2009-2010 trivalent influenza vaccine. A participant met the threshold of a 4-fold rise in titer if the Day 0 titer was less than 1:10 (the assay's lowest level of detection) and the titer at 21 days after last vaccination was 1:40 or greater, or the Day 0 titer was greater than or equal to 1:10 and the titer at 21 days after last vaccination was an increase by 4-fold or more. Day 21 after last vaccination was study Day 63 for Groups 1 and 4, and study Day 42 for Groups 2 and 3.
Time Frame: Day 0 prior to first vaccination and 21 days after last vaccination
Population: Participants who received all vaccinations and from whom blood was collected at the timepoint, all within 4 days of the window, are included. Two participants were excluded due to receipt of non-study vaccines and one due to Influenza-like illness. Analyses are as treated. This outcome restricts to age stratum.
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 29 | 30 | 30 | 25
Participants
  TIV H1 antigen | 23 | 14 | 19 | 18
  TIV H3 antigen | 25 | 18 | 25 | 23
  TIV B antigen | 10 | 7 | 4 | 4

6. Secondary Outcome: Number of Participants Age 36 Months to 9 Years With 4-fold or Greater Hemagglutination Inhibition Assay (HAI) Antibody Titer Increases Against the Virus Strains in the 2009-2010 Trivalent Influenza Vaccine (TIV) 21 Days Following the Last Vaccination
Description: as for outcome 5
Time Frame: Day 0 prior to first vaccination and Day 21 after last vaccination
Population: Participants who received all vaccinations and from whom blood was collected at the timepoint, all within 4 days of the window, are included. One participant was excluded due to receipt of non-study vaccine, 3 due to Influenza-like illness, and 1 due to H1N1 infection. Analyses are as treated. This outcome restricts to age stratum.
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 38 | 47 | 45 | 47
Participants
  TIV H1 antigen | 27 | 20 | 16 | 24
  TIV H3 antigen | 30 | 30 | 23 | 29
  TIV B antigen | 26 | 19 | 21 | 21

7. Secondary Outcome: Number of Participants Age 10 to 17 Years With 4-fold or Greater Hemagglutination Inhibition Assay (HAI) Antibody Titer Increases Against the Virus Strains in the 2009-2010 Trivalent Influenza Vaccine (TIV) 21 Days Following the Last Vaccination
Description: as for outcome 5
Time Frame: Day 0 prior to first vaccination and Day 21 after last vaccination
Population: Participants who received all vaccinations and from whom blood was collected at the timepoint, all within 4 days of the window, are included. Analyses are as treated. This outcome restricts to age stratum.
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 49 | 46 | 47 | 50
Participants
  TIV H1 antigen | 35 | 28 | 24 | 33
  TIV H3 antigen | 34 | 33 | 28 | 30
  TIV B antigen | 36 | 22 | 25 | 32

8. Secondary Outcome: Number of Participants Age 6 to Less Than 36 Months With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer of 1:40 or Greater Against the Virus Strains in the 2009-2010 Trivalent Influenza Vaccine (TIV) 21 Days Following the Last Vaccination
Description: Blood was collected from participants 21 days after the last vaccination for testing in the HAI assay against each strain in the 2009-2010 trivalent influenza vaccine. Each sample was tested according to standard operating procedures. A participant is counted if the value at the Day 63 timepoint was 1:40 or greater. Day 21 after last vaccination is study Day 63 for Groups 1 and 4, and study Day 42 for Groups 2 and 3.
Time Frame: Day 21 after last vaccination
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 29 | 30 | 30 | 25
Participants
  TIV H1 antigen | 29 | 30 | 29 | 24
  TIV H3 antigen | 29 | 30 | 29 | 25
  TIV B antigen | 10 | 9 | 8 | 5

9. Primary Outcome: Number of Participants Age 36 Months to 9 Years Reporting Solicited Subjective Systemic Reactions After the First Vaccination
Description: Participants or their parents/guardians maintained a memory aid to record daily the occurrence of systemic symptoms of feverishness, myalgia, headache, nausea and decreased general activity for 8 days after vaccination (Day 0-7) based on their interference with daily activities. Participants are counted if they were reported as experiencing the symptom at any severity on any of the 8 days.
Time Frame: Within 8 days (Day 0-7) post first vaccination
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 49 | 51 | 49 | 51
Participants
  Feverishness | 8 | 8 | 10 | 1
  Myalgia | 5 | 4 | 11 | 5
  Headache | 13 | 8 | 12 | 5
  Nausea | 8 | 4 | 6 | 4
  Decreased general activity | 12 | 6 | 14 | 5

10. Primary Outcome: Number of Participants Age 10 to 17 Years Reporting Solicited Subjective Systemic Reactions After the First Vaccination
Description: Participants or their parents/guardians maintained a memory aid to record daily the occurrence of systemic symptoms of feverishness, malaise, myalgia, headache, nausea and decreased general activity for 8 days after vaccination (Day 0-7) based on their interference with daily activities. Participants are counted if they were reported as experiencing the symptom at any severity on any of the 8 days.
Time Frame: Within 8 days (Day 0-7) post first vaccination
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 49 | 49 | 49 | 53
Participants
  Feverishness | 4 | 7 | 5 | 5
  Malaise | 14 | 13 | 10 | 11
  Myalgia | 8 | 9 | 5 | 5
  Headache | 11 | 17 | 11 | 12
  Nausea | 4 | 9 | 7 | 5
  Decreased general activity | 5 | 10 | 6 | 7

11. Primary Outcome: Number of Participants Age 6 to Less Than 36 Months Reporting Solicited Subjective Systemic Reactions After the Second Vaccination
Description: as for outcome 4
Time Frame: Within 8 days (Day 0-7) post second vaccination
Population: All participants receiving the second vaccination are included in the safety cohort. Analyses are as treated. This outcome measure is restricted to protocol-defined age stratum.
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 35 | 32 | 35 | 28
Participants
  Irritability | 11 | 15 | 13 | 11
  Decreased appetite | 5 | 5 | 3 | 7
  Lethargy | 6 | 2 | 4 | 5

12. Primary Outcome: Number of Participants Age 36 Months to 9 Years Reporting Solicited Subjective Systemic Reactions After the Second Vaccination
Description: as for outcome 9
Time Frame: Within 8 days (Day 0-7) post second vaccination
Population: as for outcome 11
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 47 | 51 | 48 | 51
Participants
  Feverishness | 2 | 3 | 4 | 2
  Myalgia | 5 | 2 | 3 | 3
  Headache | 5 | 2 | 4 | 2
  Nausea | 3 | 3 | 5 | 0
  Decreased general activity | 3 | 6 | 6 | 4

13. Primary Outcome: Number of Participants Age 10 to 17 Years Reporting Solicited Subjective Systemic Reactions After the Second Vaccination
Description: as for outcome 10
Time Frame: Within 8 days (Day 0-7) post second vaccination
Population: as for outcome 11
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 49 | 48 | 49 | 52
Participants
  Feverishness | 6 | 5 | 4 | 5
  Malaise | 9 | 9 | 4 | 2
  Myalgia | 7 | 1 | 5 | 5
  Headache | 15 | 8 | 11 | 8
  Nausea | 11 | 5 | 3 | 3
  Decreased general activity | 7 | 6 | 4 | 4

14. Primary Outcome: Number of Participants Age 6 to Less Than 36 Months Reporting Solicited Subjective Systemic Reactions After the Third Vaccination
Description: Participants' parents/guardians maintained a memory aid to record daily the occurrence of systemic symptoms of irritability, decreased appetite and lethargy for 8 days after vaccination (Day 0-7) based on their interference with daily activities. Participants are counted if they were reported as experiencing the symptom at any severity on any of the 8 days. Groups 1 and 4 only had a third vaccination day.
Time Frame: Within 8 days (Day 0-7) post third vaccination
Population: All participants receiving the third vaccination are included in the safety cohort. Analyses are as treated. This outcome measure is restricted to protocol-defined age stratum.
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 32 | 28
Participants
  Irritability | 9 | 8
  Decreased appetite | 5 | 2
  Lethargy | 6 | 2

15. Primary Outcome: Number of Participants Age 36 Months to 9 Years Reporting Solicited Subjective Systemic Reactions After the Third Vaccination
Description: Participants or their parents/guardians maintained a memory aid to record daily the occurrence of systemic symptoms of feverishness, myalgia, headache, nausea and decreased general activity for 8 days after vaccination (Day 0-7) based on their interference with daily activities. Participants are counted if they were reported as experiencing the symptom at any severity on any of the 8 days. Groups 1 and 4 only had a third vaccination day.
Time Frame: Within 8 days (Day 0-7) post third vaccination
Population: as for outcome 14
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 49 | 51
Participants
  Feverishness | 1 | 1
  Myalgia | 2 | 1
  Headache | 2 | 3
  Nausea | 1 | 1
  Decreased general activity | 3 | 2

16. Primary Outcome: Number of Participants Age 10 to 17 Years Reporting Solicited Subjective Systemic Reactions After the Third Vaccination
Description: Participants or their parents/guardians maintained a memory aid to record daily the occurrence of systemic symptoms of feverishness, malaise, myalgia, headache, nausea and decreased general activity for 8 days after vaccination (Day 0-7) based on their interference with daily activities. Participants are counted if they were reported as experiencing the symptom at any severity on any of the 8 days. Groups 1 and 4 only had a third vaccination day.
Time Frame: Within 8 days (Day 0-7) post third vaccination
Population: as for outcome 14
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 49 | 52
Participants
  Feverishness | 5 | 1
  Malaise | 8 | 4
  Myalgia | 3 | 4
  Headache | 9 | 7
  Nausea | 4 | 3
  Decreased general activity | 5 | 4

17. Primary Outcome: Number of Participants Age 6 to Less Than 36 Months Reporting Solicited Quantitative Systemic Reactions After the First Vaccination
Description: Participants' parents/guardians maintained a memory aid to record daily oral/axillary temperatures and the number of vomiting episodes, if experienced, for 8 days after vaccination (Day 0-7). Participants are counted as experiencing fever if they reported oral temperatures of 38.3 degrees Celsius or higher, or axillary temperatures of 37.8 degrees Celsius or higher, on any of the 8 days. Participants are counted as experiencing vomiting if they reported one or more episodes of vomiting on any of the 8 days.
Time Frame: Within 8 days (Day 0-7) post first vaccination
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 35 | 33 | 35 | 28
Participants
  Fever | 2 | 2 | 3 | 3
  Vomiting | 1 | 2 | 3 | 2

18. Primary Outcome: Number of Participants Age 36 Months to 9 Years Reporting Solicited Quantitative Systemic Reactions After the First Vaccination
Description: Participants or their parents/guardians maintained a memory aid to record daily oral/axillary temperatures and the number of vomiting episodes, if experienced, for 8 days after vaccination (Day 0-7). Participants are counted as experiencing fever if they reported oral temperatures of 38.3 degrees Celsius or higher, or axillary temperatures of 37.8 degrees Celsius or higher, on any of the 8 days. Participants are counted as experiencing vomiting if they reported one or more episodes of vomiting on any of the 8 days.
Time Frame: Within 8 days (Day 0-7) post first vaccination
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 49 | 51 | 49 | 51
Participants
  Fever | 4 | 1 | 5 | 1
  Vomiting | 9 | 0 | 3 | 1

19. Primary Outcome: Number of Participants Age 10 to 17 Years Reporting Solicited Quantitative Systemic Reactions After the First Vaccination
Description: as for outcome 18
Time Frame: Within 8 days (Day 0-7) post first vaccination
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 49 | 49 | 49 | 53
Participants
  Fever | 0 | 0 | 1 | 2
  Vomiting | 0 | 2 | 1 | 2

20. Primary Outcome: Number of Participants Age 6 to Less Than 36 Months Reporting Solicited Quantitative Systemic Reactions After the Second Vaccination
Description: as for outcome 17
Time Frame: Within 8 days (Day 0-7) post second vaccination
Population: All participants receiving the second vaccination are included in the safety cohort. One Group 2 participant did not report temperatures. Analyses are as treated. This outcome measure is restricted to protocol-defined age stratum.
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 35 | 32 | 35 | 28
Participants
  Fever | 3 | 1 | 4 | 1
  Vomiting | 0 | 2 | 3 | 2

21. Primary Outcome: Number of Participants Age 36 Months to 9 Years Reporting Solicited Quantitative Systemic Reactions After the Second Vaccination
Description: as for outcome 18
Time Frame: Within 8 days (Day 0-7) post second vaccination
Population: as for outcome 11
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 47 | 51 | 48 | 51
Participants
  Fever | 1 | 1 | 2 | 2
  Vomiting | 4 | 1 | 5 | 1

22. Primary Outcome: Number of Participants Age 10 to 17 Years Reporting Solicited Quantitative Systemic Reactions After the Second Vaccination
Description: as for outcome 18
Time Frame: Within 8 days (Day 0-7) post second vaccination
Population: All participants receiving the second vaccination are included in the safety cohort. One Group 3 participant did not report temperatures. Analyses are as treated. This outcome measure is restricted to protocol-defined age stratum.
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 49 | 48 | 49 | 52
Participants
  Fever | 2 | 0 | 1 | 1
  Vomiting | 3 | 1 | 1 | 2

23. Primary Outcome: Number of Participants Age 6 to Less Than 36 Months Reporting Solicited Quantitative Systemic Reactions After the Third Vaccination
Description: Participants' parents/guardians maintained a memory aid to record daily oral/axillary temperatures and the number of vomiting episodes, if experienced, for 8 days after vaccination (Day 0-7). Participants are counted as experiencing fever if they reported oral temperatures of 38.3 degrees Celsius or higher, or axillary temperatures of 37.8 degrees Celsius or higher, on any of the 8 days. Participants are counted as experiencing vomiting if they reported one or more episodes of vomiting on any of the 8 days. Groups 1 and 4 only had a third vaccination day.
Time Frame: Within 8 days (Day 0-7) post third vaccination
Population: as for outcome 14
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 32 | 28
Participants
  Fever | 3 | 2
  Vomiting | 2 | 0

24. Primary Outcome: Number of Participants Age 36 Months to 9 Years Reporting Solicited Quantitative Systemic Reactions After the Third Vaccination
Description: Participants or their parents/guardians maintained a memory aid to record daily oral/axillary temperatures and the number of vomiting episodes, if experienced, for 8 days after vaccination (Day 0-7). Participants are counted as experiencing fever if they reported oral temperatures of 38.3 degrees Celsius or higher, or axillary temperatures of 37.8 degrees Celsius or higher, on any of the 8 days. Participants are counted as experiencing vomiting if they reported one or more episodes of vomiting on any of the 8 days. Groups 1 and 4 only had a third vaccination day.
Time Frame: Within 8 days (Day 0-7) post third vaccination
Population: as for outcome 14
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 49 | 51
Participants
  Fever | 0 | 0
  Vomiting | 1 | 0

25. Primary Outcome: Number of Participants Age 10 to 17 Years Reporting Solicited Quantitative Systemic Reactions After the Third Vaccination
Description: as for outcome 24
Time Frame: Within 8 days (Day 0-7) post third vaccination
Population: as for outcome 14
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 49 | 52
Participants
  Fever | 0 | 1
  Vomiting | 0 | 1

26. Primary Outcome: Number of Participants Age 6 to Less Than 36 Months Reporting Solicited Subjective Local Reactions After the First H1N1 Vaccination
Description: Participants' parents/guardians maintained a memory aid to record daily the occurrence of local reactions of pain, tenderness and swelling for 8 days after vaccination (Day 0-7) based on their interference with daily activities. Participants are counted if they were reported as experiencing the symptom at any severity on any of the 8 days. First H1N1 vaccination was given on Study Day 0 for Groups 1, 2 and 3, and on Study Day 21 for Group 4.
Time Frame: Within 8 days (Day 0-7) post first H1N1 vaccination
Population: All participants receiving the first H1N1 vaccination are included in the safety cohort. Analyses are as treated. This outcome measure is restricted to protocol-defined age stratum.
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 35 | 33 | 35 | 28
Participants
  Pain | 1 | 6 | 8 | 1
  Tenderness | 11 | 11 | 15 | 9
  Swelling | 4 | 10 | 5 | 7

27. Primary Outcome: Number of Participants Age 36 Months to 9 Years Reporting Solicited Subjective Local Reactions After the First H1N1 Vaccination
Description: Participants or their parents/guardians maintained a memory aid to record daily the occurrence of local reactions of pain, tenderness and swelling for 8 days after vaccination (Day 0-7) based on their interference with daily activities. Participants are counted if they were reported as experiencing the symptom at any severity on any of the 8 days. First H1N1 vaccination was given on Study Day 0 for Groups 1, 2 and 3, and on Study Day 21 for Group 4.
Time Frame: Within 8 days (Day 0-7) post first H1N1 vaccination
Population: as for outcome 26
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 49 | 51 | 49 | 51
Participants
  Pain | 15 | 13 | 13 | 14
  Tenderness | 16 | 26 | 21 | 21
  Swelling | 11 | 10 | 9 | 8

28. Primary Outcome: Number of Participants Age 10 to 17 Years Reporting Solicited Subjective Local Reactions After the First H1N1 Vaccination
Description: as for outcome 27
Time Frame: Within 8 days (Day 0-7) post first H1N1 vaccination
Population: as for outcome 26
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 49 | 49 | 49 | 52
Participants
  Pain | 16 | 10 | 13 | 14
  Tenderness | 22 | 11 | 18 | 15
  Swelling | 5 | 3 | 6 | 6

29. Primary Outcome: Number of Participants Age 6 to Less Than 36 Months Reporting Solicited Subjective Local Reactions After the Second H1N1 Vaccination
Description: Participants' parents/guardians maintained a memory aid to record daily the occurrence of local reactions of pain, tenderness and swelling for 8 days after vaccination (Day 0-7) based on their interference with daily activities. Participants are counted if they were reported as experiencing the symptom at any severity on any of the 8 days. Second H1N1 vaccination was given on Study Day 21 for Groups 1, 2 and 3, and on Study Day 42 for Group 4.
Time Frame: Within 8 days (Day 0-7) post second H1N1 vaccination
Population: All participants receiving the second H1N1 vaccination are included in the safety cohort. Analyses are as treated. This outcome measure is restricted to protocol-defined age stratum.
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 35 | 32 | 35 | 28
Participants
  Pain | 4 | 5 | 10 | 1
  Tenderness | 8 | 7 | 18 | 9
  Swelling | 6 | 5 | 6 | 4

30. Primary Outcome: Number of Participants Age 36 Months to 9 Years Reporting Solicited Subjective Local Reactions After the Second H1N1 Vaccination
Description: Participants or their parents/guardians maintained a memory aid to record daily the occurrence of local reactions of pain, tenderness and swelling for 8 days after vaccination (Day 0-7) based on their interference with daily activities. Participants are counted if they were reported as experiencing the symptom at any severity on any of the 8 days. Second H1N1 vaccination was given on Study Day 21 for Groups 1, 2 and 3, and on Study Day 42 for Group 4.
Time Frame: Within 8 days (Day 0-7) post second H1N1 vaccination
Population: as for outcome 29
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 47 | 51 | 48 | 51
Participants
  Pain | 16 | 14 | 17 | 10
  Tenderness | 20 | 23 | 20 | 21
  Swelling | 8 | 8 | 9 | 9

31. Primary Outcome: Number of Participants Age 10 to 17 Years Reporting Solicited Subjective Local Reactions After the Second H1N1 Vaccination
Description: as for outcome 30
Time Frame: Within 8 days (Day 0-7) post second H1N1 vaccination
Population: as for outcome 29
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 49 | 48 | 49 | 52
Participants
  Pain | 16 | 14 | 19 | 7
  Tenderness | 22 | 16 | 23 | 15
  Swelling | 4 | 5 | 9 | 4

32. Primary Outcome: Number of Participants Age 6 to Less Than 36 Months Reporting Solicited Subjective Local Reactions After the TIV Vaccination
Description: Participants' parents/guardians maintained a memory aid to record daily the occurrence of local reactions of pain, tenderness and swelling for 8 days after vaccination (Day 0-7) based on their interference with daily activities. Participants are counted if they were reported as experiencing the symptom at any severity on any of the 8 days. The TIV vaccination was given on Study Day 42 for Group 1, Study Day 0 for Groups 2 and 4, and on Study Day 21 for Group 3.
Time Frame: Within 8 days (Day 0-7) post TIV vaccination
Population: All participants receiving the TIV vaccination are included in the safety cohort. Analyses are as treated. This outcome measure is restricted to protocol-defined age stratum.
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 32 | 33 | 35 | 28
Participants
  Pain | 3 | 6 | 7 | 1
  Tenderness | 8 | 10 | 15 | 5
  Swelling | 6 | 9 | 7 | 7

33. Primary Outcome: Number of Participants Age 36 Months to 9 Years Reporting Solicited Subjective Local Reactions After the TIV Vaccination
Description: Participants or their parents/guardians maintained a memory aid to record daily the occurrence of local reactions of pain, tenderness and swelling for 8 days after vaccination (Day 0-7) based on their interference with daily activities. Participants are counted if they were reported as experiencing the symptom at any severity on any of the 8 days. The TIV vaccination was given on Study Day 42 for Group 1, Study Day 0 for Groups 2 and 4, and on Study Day 21 for Group 3.
Time Frame: Within 8 days (Day 0-7) post TIV vaccination
Population: as for outcome 32
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 49 | 51 | 48 | 51
Participants
  Pain | 21 | 14 | 20 | 24
  Tenderness | 21 | 23 | 23 | 30
  Swelling | 7 | 8 | 8 | 16

34. Primary Outcome: Number of Participants Age 10 to 17 Years Reporting Solicited Subjective Local Reactions After the TIV Vaccination
Description: as for outcome 33
Time Frame: Within 8 days (Day 0-7) post TIV vaccination
Population: as for outcome 32
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 49 | 49 | 49 | 53
Participants
  Pain | 25 | 27 | 26 | 26
  Tenderness | 27 | 28 | 32 | 34
  Swelling | 4 | 8 | 9 | 11

35. Primary Outcome: Number of Participants Age 6 to Less Than 36 Months Reporting Solicited Quantitative Local Reactions After the First H1N1 Vaccination
Description: Participants' parents/guardians maintained a memory aid to record daily the occurrence of local reactions of swelling and redness for 8 days (Day 0-7) after vaccination. If the reaction was present, the maximum diameter was measured in millimeters (mm). Participants are counted if they were reported as experiencing the reaction with any measurement greater than 0 mm on any of the 8 days. First H1N1 vaccination was given on Study Day 0 for Groups 1, 2 and 3, and on Study Day 21 for Group 4.
Time Frame: Within 8 days (Day 0-7) post first H1N1 vaccination
Population: as for outcome 26
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 35 | 33 | 35 | 28
Participants
  Redness | 14 | 15 | 15 | 17
  Swelling | 4 | 10 | 5 | 9

36. Primary Outcome: Number of Participants Age 36 Months to 9 Years Reporting Solicited Quantitative Local Reactions After the First H1N1 Vaccination
Description: Participants or their parents/guardians maintained a memory aid to record daily the occurrence of local reactions of swelling and redness for 8 days (Day 0-7) after vaccination. If the reaction was present, the maximum diameter was measured in millimeters (mm). Participants are counted if they reported experiencing the reaction with any measurement greater than 0 mm on any of the 8 days. First H1N1 vaccination was given on Study Day 0 for Groups 1, 2 and 3, and on Study Day 21 for Group 4.
Time Frame: Within 8 days (Day 0-7) post first H1N1 vaccination
Population: as for outcome 26
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 49 | 51 | 49 | 51
Participants
  Redness | 19 | 18 | 23 | 16
  Swelling | 12 | 12 | 9 | 8

37. Primary Outcome: Number of Participants Age 10 to 17 Years Reporting Solicited Quantitative Local Reactions After the First H1N1 Vaccination
Description: as for outcome 36
Time Frame: Within 8 days (Day 0-7) post first H1N1 vaccination
Population: as for outcome 26
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 49 | 49 | 49 | 52
Participants
  Redness | 8 | 6 | 15 | 14
  Swelling | 6 | 4 | 6 | 6

38. Primary Outcome: Number of Participants Age 6 to Less Than 36 Months Reporting Solicited Quantitative Local Reactions After the Second H1N1 Vaccination
Description: Participants' parents/guardians maintained a memory aid to record daily the occurrence of local reactions of swelling and redness for 8 days (Day 0-7) after vaccination. If the reaction was present, the maximum diameter was measured in millimeters (mm). Participants are counted if they were reported as experiencing the reaction with any measurement greater than 0 mm on any of the 8 days. Second H1N1 vaccination was given on Study Day 21 for Groups 1, 2 and 3, and on Study Day 42 for Group 4.
Time Frame: Within 8 days (Day 0-7) post second H1N1 vaccination
Population: as for outcome 29
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 35 | 32 | 35 | 28
Participants
  Redness | 14 | 17 | 14 | 14
  Swelling | 7 | 8 | 9 | 5

39. Primary Outcome: Number of Participants Age 36 Months to 9 Years Reporting Solicited Quantitative Local Reactions After the Second H1N1 Vaccination
Description: Participants or their parents/guardians maintained a memory aid to record daily the occurrence of local reactions of swelling and redness for 8 days (Day 0-7) after vaccination. If the reaction was present, the maximum diameter was measured in millimeters (mm). Participants are counted if they reported experiencing the reaction with any measurement greater than 0 mm on any of the 8 days. Second H1N1 vaccination was given on Study Day 21 for Groups 1, 2 and 3, and on Study Day 42 for Group 4.
Time Frame: Within 8 days (Day 0-7) post second H1N1 vaccination
Population: as for outcome 29
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 47 | 51 | 48 | 51
Participants
  Redness | 12 | 19 | 22 | 18
  Swelling | 8 | 9 | 11 | 10

40. Primary Outcome: Number of Participants Age 10 to 17 Years Reporting Solicited Quantitative Local Reactions After the Second H1N1 Vaccination
Description: as for outcome 39
Time Frame: Within 8 days (Day 0-7) post second H1N1 vaccination
Population: as for outcome 29
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 49 | 48 | 49 | 52
Participants
  Redness | 15 | 13 | 14 | 13
  Swelling | 5 | 5 | 9 | 4

41. Primary Outcome: Number of Participants Age 6 to Less Than 36 Months Reporting Solicited Quantitative Local Reactions After the TIV Vaccination
Description: Participants' parents/guardians maintained a memory aid to record daily the occurrence of local reactions of swelling and redness for 8 days (Day 0-7) after vaccination. If the reaction was present, the maximum diameter was measured in millimeters (mm). Participants are counted if they were reported as experiencing the reaction with any measurement greater than 0 mm on any of the 8 days. The TIV vaccination was given on Study Day 42 for Group 1, Study Day 0 for Groups 2 and 4, and on Study Day 21 for Group 3.
Time Frame: Within 8 days (Day 0-7) post TIV vaccination
Population: as for outcome 32
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 32 | 33 | 35 | 28
Participants
  Redness | 17 | 14 | 16 | 17
  Swelling | 6 | 9 | 9 | 9

42. Primary Outcome: Number of Participants Age 36 Months to 9 Years Reporting Solicited Quantitative Local Reactions After the TIV Vaccination
Description: Participants or their parents/guardians maintained a memory aid to record daily the occurrence of local reactions of swelling and redness for 8 days (Day 0-7) after vaccination. If the reaction was present, the maximum diameter was measured in millimeters (mm). Participants are counted if they reported experiencing the reaction with any measurement greater than 0 mm on any of the 8 days. The TIV vaccination was given on Study Day 42 for Group 1, Study Day 0 for Groups 2 and 4, and on Study Day 21 for Group 3.
Time Frame: Within 8 days (Day 0-7) post TIV vaccination
Population: as for outcome 32
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 49 | 51 | 48 | 51
Participants
  Redness | 16 | 19 | 20 | 18
  Swelling | 8 | 14 | 10 | 10

43. Primary Outcome: Number of Participants Age 10 to 17 Years Reporting Solicited Quantitative Local Reactions After the TIV Vaccination
Description: as for outcome 42
Time Frame: Within 8 days (Day 0-7) post TIV vaccination
Population: as for outcome 32
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 49 | 49 | 49 | 53
Participants
  Redness | 15 | 10 | 15 | 15
  Swelling | 4 | 8 | 9 | 11

44. Primary Outcome: Number of Participants Reporting Vaccine-associated Serious Adverse Events (SAEs)
Description: Serious adverse events included any untoward medical occurrence that resulted in death; was life threatening; was a persistent/significant disability/incapacity; required in-patient hospitalization or prolongation thereof; resulted in a congenital anomaly/birth defect; may have jeopardized the participant or required intervention to prevent one of these outcomes; or was described as Guillain-Barré Syndrome. Association to vaccination was determined by a study clinician licensed to make medical diagnoses.
Time Frame: Day 0 through 180 days after the last vaccination
Population: All participants receiving at least one vaccination are included in the safety cohort. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 133 | 133 | 133 | 132
Participants | 0 | 0 | 0 | 0

45. Primary Outcome: Number of Participants Age 6 Months to Less Than 36 Months With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer of 1:40 or Greater Against the H1N1 2009 Virus 21 Days Following the First Dose of H1N1 Vaccine
Description: Blood was collected from all participants 21 days after vaccination for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. For Group 4, this timepoint is Study Day 42, all others it is Study Day 21. Each sample was tested at least twice according to standard operating procedures and the result of each replicate reported. A participant is counted if the geometric mean of the replicate values was 1:40 or greater.
Time Frame: Day 21 after first H1N1 vaccination
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 35 | 32 | 33 | 26
Participants | 10 | 6 | 5 | 5

46. Primary Outcome: Number of Participants Age 36 Months to 9 Years With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer of 1:40 or Greater Against the H1N1 2009 Virus 21 Days Following the First Dose of H1N1 Vaccine
Description: as for outcome 45
Time Frame: Day 21 after first H1N1 vaccination
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 47 | 49 | 45 | 50
Participants | 20 | 21 | 19 | 22

47. Primary Outcome: Number of Participants Age 10 to 17 Years With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer of 1:40 or Greater Against the H1N1 2009 Virus 21 Days Following the First Dose of H1N1 Vaccine
Description: as for outcome 45
Time Frame: Day 21 after first H1N1 vaccination
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 49 | 48 | 46 | 51
Participants | 47 | 40 | 45 | 48

48. Secondary Outcome: Number of Participants Age 36 Months to 9 Years With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer of 1:40 or Greater Against the Virus Strains in the 2009-2010 Trivalent Influenza Vaccine (TIV) 21 Days Following the Last Vaccination
Description: as for outcome 8
Time Frame: Day 21 after last vaccination
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 38 | 47 | 45 | 47
Participants
  TIV H1 antigen | 38 | 43 | 44 | 47
  TIV H3 antigen | 38 | 43 | 44 | 47
  TIV B antigen | 32 | 31 | 33 | 34

49. Secondary Outcome: Number of Participants Age 10 to 17 Years With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer of 1:40 or Greater Against the Virus Strains in the 2009-2010 Trivalent Influenza Vaccine (TIV) 21 Days Following the Last Vaccination
Description: as for outcome 8
Time Frame: Day 21 after last vaccination
Population: as for outcome 7
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 49 | 46 | 47 | 50
Participants
  TIV H1 antigen | 49 | 46 | 46 | 50
  TIV H3 antigen | 49 | 46 | 46 | 50
  TIV B antigen | 47 | 35 | 40 | 47

50. Secondary Outcome: Number of Participants Age 6 to Less Than 36 Months With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer of 1:40 or Greater Against the H1N1 2009 Virus 21 Days Following the Second Dose of H1N1 Vaccine
Description: Blood was collected from all participants 21 days after vaccination for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. For Group 4, 21 days after second H1N1 vaccination is study Day 63, all others it is study Day 42. Each sample was tested at least twice according to standard operating procedures and the result of each replicate reported. A participant is counted if the geometric mean of the replicate values was 1:40 or greater.
Time Frame: Day 21 after the second H1N1 vaccination
Population: Participants who received all vaccinations and from whom blood was collected at the timepoint, all within 4 days of the window, are included. One participant was excluded due to receipt of a non-study vaccine and one due to Influenza-like illness. Analyses are as treated. This outcome restricts to age stratum.
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 30 | 31 | 31 | 26
Participants | 23 | 24 | 26 | 19

51. Secondary Outcome: Number of Participants Age 36 Months to 9 Years With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer of 1:40 or Greater Against the H1N1 2009 Virus 21 Days Following the Second Dose of H1N1 Vaccine
Description: as for outcome 50
Time Frame: Day 21 after the second H1N1 vaccination
Population: as for outcome 50
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 44 | 47 | 45 | 47
Participants | 38 | 37 | 36 | 37

52. Secondary Outcome: Number of Participants Age 10 to 17 Years With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer of 1:40 or Greater Against the H1N1 2009 Virus 21 Days Following the Second Dose of H1N1 Vaccine
Description: as for outcome 50
Time Frame: Day 21 after the second H1N1 vaccination
Population: Participants who received all vaccinations and from whom blood was collected at the timepoint, all within 4 days of the window, are included. This outcome restricts to age stratum.
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 49 | 46 | 47 | 50
Participants | 49 | 42 | 47 | 50

53. Secondary Outcome: Number of Participants Age 6 to Less Than 36 Months With 4-fold or Greater Hemagglutination Inhibition Assay (HAI) Antibody Titer Increases Against the Influenza H1N1 2009 Virus 21 Days Following the Second Dose of H1N1 Vaccine
Description: Blood was collected from participants for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. A participant met the threshold of a 4-fold rise in titer if the Day 0 titer was less than 1:10 (the assay's lowest level of detection) and the Day 21 post second H1N1 vaccination titer was 1:40 or greater, or the Day 0 titer was greater than or equal to 1:10 and the Day 21 titer was an increase by 4-fold or more. Day 21 post second H1N1 vaccination is study Day 63 for Group 4, and is study Day 42 for all other groups.
Time Frame: Day 0 prior to first vaccination and 21 days after the second H1N1 vaccination
Population: as for outcome 50
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 30 | 30 | 31 | 26
Participants | 23 | 23 | 26 | 19

54. Secondary Outcome: Number of Participants Age 36 Months to 9 Years With 4-fold or Greater Hemagglutination Inhibition Assay (HAI) Antibody Titer Increases Against the Influenza H1N1 2009 Virus 21 Days Following the Second Dose of H1N1 Vaccine
Description: as for outcome 53
Time Frame: Day 0 prior to first vaccination and 21 days after the second H1N1 vaccination
Population: as for outcome 50
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 44 | 47 | 45 | 47
Participants | 38 | 37 | 36 | 35

55. Secondary Outcome: Number of Participants Age 10 to 17 Years With 4-fold or Greater Hemagglutination Inhibition Assay (HAI) Antibody Titer Increases Against the Influenza H1N1 2009 Virus 21 Days Following the Second Dose of H1N1 Vaccine
Description: as for outcome 53
Time Frame: Day 0 prior to first vaccination and 21 days after the second H1N1 vaccination
Population: as for outcome 7
Measure: Number; unit: Participants
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Number analyzed (Participants) | 49 | 46 | 47 | 50
Participants | 48 | 41 | 43 | 50

ADVERSE EVENTS:
Time Frame: Solicited events were collected for 8 days after each vaccination, unsolicited events through 21 days after last vaccination, and serious adverse events and new onset chronic medical conditions through 180 days after last vaccination.
Description: For events solicited on a Memory Aid in the 8 days after vaccination, a participant was considered to have one event if it was reported as experienced at any time in the 8 day period.
Arm/Group | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 | Group 3: Day 0-H1N1; Day 21-H1N1+TIV | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1
Serious Adverse Events (participants affected / at risk) | 0/133 | 3/133 | 1/133 | 2/132
Other Adverse Events (participants affected / at risk) | 124/133 | 125/133 | 124/133 | 125/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV (N=133) | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 (N=133) | Group 3: Day 0-H1N1; Day 21-H1N1+TIV (N=133) | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1 (N=132)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Group 1: Day 0-H1N1; Day 21-H1N1; Day 42-TIV (N=133) | Group 2: Day 0-H1N1+TIV; Day 21-H1N1 (N=133) | Group 3: Day 0-H1N1; Day 21-H1N1+TIV (N=133) | Group 4: Day 0-TIV; Day 21-H1N1; Day 42-H1N1 (N=132)
Cough (Respiratory, thoracic and mediastinal disorders) | 16 (16) | 9 (10) | 9 (10) | 21 (23)
Diarrhoea (Gastrointestinal disorders) | 18 (22) | 6 (7) | 9 (13) | 10 (13)
Injection site haematoma (General disorders) | 3 (3) | 8 (9) | 6 (6) | 4 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 11 (11) | 8 (8) | 11 (11)
Nasopharyngitis (Infections and infestations) | 13 (14) | 13 (14) | 10 (11) | 11 (12)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 12 (13) | 5 (5) | 4 (4) | 9 (10)
Pyrexia (General disorders) | 5 (5) | 4 (4) | 3 (3) | 8 (8)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 23 (25) | 11 (12) | 7 (7) | 12 (18)
Upper respiratory tract infection (Infections and infestations) | 16 (16) | 11 (11) | 15 (18) | 14 (20)
Pyrexia (General disorders) | 14 (15) | 5 (8) | 15 (23) | 13 (13)
Irritability (General disorders) | 22/35 (38) | 20/33 (45) | 23/35 (42) | 17/28 (28) — Solicited from participants aged 6 to less than 36 months only.
Decreased Appetite (Metabolism and nutrition disorders) | 9/35 (16) | 8/33 (15) | 11/35 (15) | 13/28 (14) — Solicited from participants aged 6 to less than 36 months only.
Lethargy (Nervous system disorders) | 14/35 (20) | 7/33 (14) | 10/35 (16) | 9/28 (10) — Solicited from participants aged 6 to less than 36 months only.
Feeling hot (General disorders) | 25/98 (26) | 21/100 (38) | 20/98 (31) | 15/104 (15) — Solicited from participants aged 36 months to 17 years only.
Malaise (General disorders) | 24/49 (31) | 15/49 (35) | 13/49 (18) | 14/53 (17) — Solicited from participants aged 10 to 17 years only.
Myalgia (Musculoskeletal and connective tissue disorders) | 21/98 (30) | 15/100 (29) | 23/98 (32) | 19/104 (23) — Solicited from participants aged 36 months to 17 years only.
Headache (Nervous system disorders) | 40/98 (55) | 27/100 (60) | 33/98 (53) | 27/104 (37) — Solicited from participants aged 36 months to 17 years only.
Nausea (Gastrointestinal disorders) | 25/98 (31) | 18/100 (34) | 19/98 (29) | 13/104 (16) — Solicited from participants aged 36 months to 17 years only.
Decreased activity (General disorders) | 27/98 (35) | 21/100 (44) | 26/98 (40) | 21/104 (26) — Solicited from participants aged 36 months to 17 years only.
Vomiting (Gastrointestinal disorders) | 16 (20) | 8 (12) | 14 (25) | 11 (11)
Injection site pain (General disorders) | 70 (117) | 67 (112) | 75 (133) | 65 (98)
Tenderness (General disorders) | 83 (155) | 82 (158) | 91 (185) | 90 (159) — Tenderness was solicited as a reaction at the vaccination site.
Injection site erythema (General disorders) | 75 (130) | 68 (131) | 76 (154) | 72 (141)
Injection site swelling (functional grading) (General disorders) | 35 (55) | 39 (70) | 39 (68) | 51 (72) — Injection site swelling was solicited separately for functional grading of impact on daily activities and as a measured reaction.
Injection site swelling (measured) (General disorders) | 37 (60) | 45 (79) | 43 (77) | 53 (77) — Injection site swelling was solicited separately for functional grading of impact on daily activities and as a measured reaction.

LIMITATIONS AND CAVEATS:
Due to difficulties identifying children in the youngest age stratum who were previously primed, enrollment in this stratum was closed prior to meeting the planned number of participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less